CLINICAL TRIAL: NCT02505607
Title: Overactive Bladder Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility issues
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Katie Propst, Fellow, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HHC-2015-0109
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Urinary Bladder, Overactive; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care Group (No Intervention): In this group, subjects will receive standard counseling regarding Overactive Bladder.
- Care Plan Group (Experimental): In this group, subjects will receive counseling regarding Overactive Bladder using a printed "Overactive Bladder Plan of Care" information sheet.
  Interventions: Other: Overactive Bladder Care Plan counseling

INTERVENTIONS:
Other: Overactive Bladder Care Plan counseling — Use of a printed "Overactive Bladder Plan of Care" information sheet.
  Arms: Care Plan Group

SUMMARY:
Overactive bladder (OAB) is a common, chronic condition, characterized by urinary "urgency, with or without urge incontinence, usually with frequency and nocturia." Treatment adherence is a major barrier to management of OAB and drug continuation is poor. Many factors may play a role in non-adherence to medication management of OAB including drug cost, side effects, and a lack of understanding of the disease and treatment process.Studies show that recall of disease information and treatment is often suboptimal. Literature shows that providing written materials is an efficacious way to aid in recall. Based on known poor adherence to OAB medication treatment and the clear role patient education methods have on patient information recall, the investigators believe that improvement of participant education through use of a OAB care plan will improve participant understanding and treatment adherence.

Through this randomized trial, the investigators plan to evaluate whether implementation of a OAB Care Plan improves understanding of disease and treatment options, treatment success, and satisfaction.

This is a prospective, randomized, controlled study of OAB counseling in new patients presenting to the Urogynecology offices of Hartford Hospital. All new patients with a diagnosis of OAB will be offered participation. All consenting participants will be randomized 1:1 to one of two groups: 1) Standard Care group or 2) Care Plan group. In the Standard Care group, participants will be counseled as the physician routinely counsels patients about OAB, in the Care Plan group, participants will be counseled a printed "Overactive Bladder Plan of Care" information sheet. At the end of the visit, the participant will complete a Baseline Survey. The Baseline Survey includes basic demographic information, a physician satisfaction survey, and a OAB knowledge survey. The participant will return for follow up as directed by the physician.

At the follow up visit, participants in both groups will complete a Followup Survey. The Followup Survey will be completed before the participant sees the physician. The Followup Survey assesses OAB knowledge.

Eight months after the baseline visit, each participant's chart will be reviewed for final data collection. If a participant progresses to a treatment method where she is satisfied and would like to remain, this will be documented.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of overactive bladder
* able and willing to participate and consent
* age >17 years, <90 years
* female sex

Exclusion Criteria:

* male sex
* patients who do not have a diagnosis of overactive bladder
* age <18 years, >89 years
* unable or unwilling to participate
* patients who are already being treated for overactive bladder
* patients who are planning surgical intervention for pelvic organ prolapse prior to treatment of overactive bladder
* patients who are planning surgical intervention for stress urinary incontinence prior to treatment of overactive bladder
* pregnancy

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Understanding of Overactive Bladder questionnaire | Change from baseline knowledge at follow up visit (on average 8 weeks)

SECONDARY OUTCOMES:
Subject satisfaction questionnaire | Baseline visit (time 0)
Treatment success chart review | 8 months after baseline visit

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hartford Hospital, Urogynecology Division, Glastonbury, Connecticut
  - Hartford Hospital, Urogynecology Division, Hartford, Connecticut
  - Hartford Hospital, Urogynecology Division, West Hartford, Connecticut

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] D'Souza AO, Smith MJ, Miller LA, Doyle J, Ariely R. Persistence, adherence, and switch rates among extended-release and immediate-release overactive bladder medications in a regional managed care plan. J Manag Care Pharm. 2008 Apr;14(3):291-301. doi: 10.18553/jmcp.2008.14.3.291. PMID 18439051
- [Background] Yeaw J, Benner JS, Walt JG, Sian S, Smith DB. Comparing adherence and persistence across 6 chronic medication classes. J Manag Care Pharm. 2009 Nov-Dec;15(9):728-40. doi: 10.18553/jmcp.2009.15.9.728. PMID 19954264
- [Background] Pickney CS, Arnason JA. Correlation between patient recall of bone densitometry results and subsequent treatment adherence. Osteoporos Int. 2005 Sep;16(9):1156-60. doi: 10.1007/s00198-004-1818-8. Epub 2005 Mar 3. PMID 15744452
- [Background] Watson PW, McKinstry B. A systematic review of interventions to improve recall of medical advice in healthcare consultations. J R Soc Med. 2009 Jun;102(6):235-43. doi: 10.1258/jrsm.2009.090013. PMID 19531618